CLINICAL TRIAL: NCT06113445
Title: A Phase 3, Randomized, Double-Blind, 52-Week, Placebo-Controlled, Efficacy and Safety Study of Povorcitinib in Participants With Nonsegmental Vitiligo
Brief Title: A Study to Evaluate Efficacy and Safety of Povorcitinib in Participants With Nonsegmental Vitiligo (STOP-V1)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB54707-303; 2023-505782-86-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: NonSegmental Vitiligo

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: Povorcitinib Dose A (Experimental): Participants will receive Povorcitinib Dose A for 52 weeks, followed by Povorcitinib Dose A for 52 weeks.
  Interventions: Drug: Povorcitinib
- Placebo (Placebo Comparator): Participants will receive Placebo for 52 weeks, followed by Povorcitinib Dose A for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Povorcitinib — Oral, Tablet
  Other Names: INCB054707
  Arms: Experimental: Povorcitinib Dose A
Drug: Placebo — Oral, Tablet
  Arms: Placebo

SUMMARY:
This study is being conducted to determine the efficacy and safety of povorcitinib in participants with nonsegmental vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years.
* Clinical diagnosis of nonsegmental vitiligo and meet the following:

  * T-BSA ≥ 5%
  * T-VASI score ≥ 4
  * F-BSA ≥ 0.5%
  * F-VASI score ≥ 0.5
* Agreement to discontinue all agents and procedures used to treat vitiligo from screening through the final safety follow-up visit.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Other forms of vitiligo or skin depigmentation disorders.
* Clinically significant abnormal TSH or free T4 at screening.
* Use of laser or phototherapy within 8 weeks and dihydroxyacetone within 4 weeks prior to Day 1.
* Current or past use of the depigmenting agent monobenzyl ether of hydroquinone including Benoquin®.
* History of melanocyte-keratinocyte transplantation procedure or other surgical treatment for vitiligo.
* Spontaneous and significant repigmentation within 6 months prior to screening.
* Women who are pregnant, considering pregnancy, or breast feeding.
* Medical history including thrombocytopenia, coagulopathy or platelet dysfunction; venous and arterial thrombosis, deep vein thrombosis, pulmonary embolism, stroke, moderate to severe heart failure, cerebrovascular accident, myocardial infarction, or other significant cardiovascular diseases; Q-wave interval abnormalities; disseminated herpes zoster or recurrent dermatomal herpes zoster; disseminated herpes simplex; chronic/recurrent infections; malignancies.
* Evidence of infection with TB, HBV, HCV or HIV.
* History of failure to JAK inhibitor treatment of any inflammatory disease.
* Laboratory values outside of the protocol-defined ranges.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2027-02-24 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving a ≥ 75% Improvement From Baseline in the Facial Vitiligo Area Scoring Index (F-VASI75) | Week 52
  ≥75% improvement in facial Vitiligo Area Scoring Index.

SECONDARY OUTCOMES:
Percentage change from Baseline in Total Body Vitiligo Area Scoring Index (T-VASI) | Week 52
  Percentage change from Baseline in total body Vitiligo Area Scoring Index.
Proportion of Participants Achieving a ≥ 50% Improvement From Baseline in the Total Body Vitiligo Area Scoring Index (T-VASI50) | Week 52
  ≥50% improvement in total body Vitiligo Area Scoring Index.
Proportion of Participants Achieving a ≥ 75% Improvement From Baseline in the Total Body Vitiligo Area Scoring Index (T-VASI75) | Week 52
  ≥75% improvement in total body Vitiligo Area Scoring Index
Proportion of participants achieving a Vitiligo Noticeability Scale Score (VNS) of 4 or 5 | Week 52 and Week 104
  VNS is a participant reported outcome measure on a scale of 1-5, 1- more noticeable, 4 - a lot less noticeable, and 5- no longer noticeable.
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to Week 104 and 30 days
  Defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug.
Proportion of Participants Achieving Facial Vitiligo Area Scoring Index (F-VASI50) | Week 52 and Week 104
  ≥50% improvement in facial Vitiligo Area Scoring Index.
Proportion of Participants Achieving Facial Vitiligo Area Scoring Index (F-VASI75) | Week 104
  ≥75% improvement in facial Vitiligo Area Scoring Index.
Proportion of Participants Achieving Facial Vitiligo Area Scoring Index (F-VASI90) | Week 52 and Week 104
  ≥90% improvement in facial Vitiligo Area Scoring Index.
Proportion of Participants Achieving Total Body Vitiligo Area Scoring Index (T-VASI50) | Week 104
  ≥50% improvement in total body Vitiligo Area Scoring Index.
Proportion of Participants Achieving Total Body Vitiligo Area Scoring Index (T-VASI75) | Week 104
  ≥75% improvement in total body Vitiligo Area Scoring Index.
Proportion of Participants Achieving Total Body Vitiligo Area Scoring Index (T-VASI90) | Week 52 and Week 104
  ≥90% improvement in total body Vitiligo Area Scoring Index.
Proportion of participants achieving an Facial Static Investigator Global Assessment (FSIGA) of 0 or 1 | Week 52 and Week 104
  Global score of vitiligo severity for the face. Scores range from 0 (clear) to 5 (severe vitiligo).
Proportion of participants in each Facial Static Investigator Global Assessment (FSIGA) category | Week 52 and Week 104
  Global score of vitiligo severity for the face. Scores range from 0 (clear) to 5 (severe vitiligo).
Proportion of participants achieving a Static Investigator Global Assessment (SIGA) of 0 (clear) or 1 (almost clear) | Week 52 and Week 104
  Global score of vitiligo severity for the entire body. Scores range from 0 (clear) to 5 (severe vitiligo).
Proportion of participants in each Static Investigator Global Assessment (SIGA) category | Week 52 and Week 104
  Global score of vitiligo severity for the entire body. Scores range from 0 (clear) to 5 (severe vitiligo).
Proportion of participants who report Facial Patient Global Impression of Change-Vitiligo (F-PaGIC-V) of 1 or 2 | Week 52 and Week 104
  F-PaGIC-V is an assessment of improvement of vitiligo on the face by the participant. It is a 7-point scale ((1) Very much improved, (2) Much improved, (3) Minimally improved, (4) No change, (5) Minimally worse, (6) Much worse, or (7) Very much worse).
Proportion of participants in each Facial Patient Global Impression of Change-Vitiligo (F-PaGIC-V) category | Week 52 and Week 104
  F-PaGIC-V is an assessment of improvement of vitiligo on the face by the participant. It is a 7-point scale ((1) Very much improved, (2) Much improved, (3) Minimally improved, (4) No change, (5) Minimally worse, (6) Much worse, or (7) Very much worse).
Proportion of participants who report Total Body Patient Global Impression of Change-Vitiligo (T-PaGIC-V) of 1 or 2 | Week 52 and Week 104
  T-PaGIC-V is an assessment of improvement of vitiligo on the total body by the participant. It is a 7-point scale ((1) Very much improved, (2) Much improved, (3) Minimally improved, (4) No change, (5) Minimally worse, (6) Much worse, or (7) Very much worse).
Proportion of participants in each Total Body Patient Global Impression of Change-Vitiligo (T-PaGIC-V) category | Week 52 and Week 104
  T-PaGIC-V is an assessment of improvement of vitiligo on the total body by the participant. It is a 7-point scale ((1) Very much improved, (2) Much improved, (3) Minimally improved, (4) No change, (5) Minimally worse, (6) Much worse, or (7) Very much worse).
Proportion of participants in each category for the color-matching question | Week 52 and Week 104
  Participants will answer how well the color of the treated skin matches the normal skin on a scale of 1-5, 1 being excellent to 5 being very poor.
Change from baseline in the Vitiligo-Specific Quality of Life (VitiQoL) | Week 52 and Week 104
  VitiQoL is a 15-item QoL assessment that asks participants to rate various aspects of their condition during the past month using a 7-point scale ("Not at all" to "All of the time").
Change from baseline in the Hospital Anxiety and Depression Scale (HADS) subscales | Week 52 and Week 104
  HADS is a 14-item questionnaire that assesses the levels of anxiety and depression that a participant is currently experiencing. There are 7 questions each for measuring anxiety and for measuring depression, with 4 possible responses to each question (responses are scored as 0, 1, 2, or 3).

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (100):
- United States (34):
  - Cahaba Dermatology, Hoover, Alabama
  - University of California Irvine, Irvine, California
  - Clinical Science Institute Clinical Research Specialists Inc, Santa Monica, California
  - Cura Clinical Research, Sherman Oaks, California
  - Sutter Health Palo Alto Medical Foundation Pamf Sunnyvale Center, Sunnyvale, California
  - Renaissance Research, Cape Coral, Florida
  - Encore Medical Research, Llc, Hollywood, Florida
  - Savin Medical Group, Rc, Miami, Florida
  - Skin Research of South Florida, Llc, Miami, Florida
  - San Marcus Research Clinic Inc., Miami Lakes, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Forcare Clinical Research, Tampa, Florida
  - Cleaver Medical Group, Cumming, Georgia
  - Dermatology and Surgery Specialists of North Atlanta, Marietta, Georgia
  - Pivotal Research Solutions, Stonecrest, Georgia
  - Options Research Group, Llc, Kokomo, Indiana
  - Allcutis Research, Llc, Beverly, Massachusetts
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - Great Lakes Research Group Inc, Bay City, Michigan
  - Wayne State University Physician Group Dermatology, Dearborn, Michigan
  - Revival Research Institute, Llc Dermatology, Troy, Michigan
  - Medisearch Clinical Trials, Saint Joseph, Missouri
  - Jdr Dermatology Research, Las Vegas, Nevada
  - Empire Dermatology, East Syracuse, New York
  - Sadick Dermatology Sadick Research Group, New York, New York
  - Derm Research Center of New York Inc, Stony Brook, New York
  - Dermatology Associates of Plymouth Meeting, Plymouth Meeting, Pennsylvania
  - International Clinical Research Tennessee Llc, Murfreesboro, Tennessee
  - University of Texas Physicians - Bellaire Station, Bellaire, Texas
  - Center For Clinical Studies, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Jordan Valley Dermatology Center, West Jordan, Utah
  - Clinical Research Partners Llc Crp Richmond Forest Avenue Office Building Location, Richmond, Virginia
  - Dermatology Specialists of Spokane, Spokane, Washington
- Belgium (4):
  - Hopital Universitaire de Bruxelles/ Academisch Ziekenhuis Burssel, Brussel/ Brussels/bruxelles
  - Universitair Ziekenhuis Gent (Uz Gent), Ghent
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
  - Cliniques Universitaires Ucl Saint-Luc, Woluwe-Saint-Lambert
- Canada (9):
  - Dermatology Research Institute, Calgary, Alberta
  - Enverus Medical Research, Surrey, British Columbia
  - Leader Research, Burlington, Ontario
  - Dermeffects, London, Ontario
  - North York Research Inc., North YORK, Ontario
  - Care Clinic, Ottawa, Ontario
  - Siena Medical Research Corporation, Ottawa, Ontario
  - Skin Health, Peterborough, Ontario
  - Alliance Clinical Trials, Waterloo, Ontario
- France (4):
  - Centre Hospitalier Universitaire (Chu) - Hopital Henri Mondor, Bordeaux
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Saint - Andre, Bordeaux
  - Clinique de Courlancy, Reims
  - Hopital Larrey, Toulouse
- Germany (5):
  - Universitatsklinikum Erlangen, Erlangen
  - Klinikum Der Johann Wolfgang Goethe University, Frankfurt am Main
  - Derma-Study-Center Friedrichshafen Gmbh, Friedrichshafen
  - Dermatologische Gemeinschaftspraxis Dres. Quist, Mainz
  - Beldio Research Gmbh, Memmingen
- Japan (17):
  - Hamamatsu University Hospital, Hamamatsu
  - St. Marianna University School of Medicine Hospital, Kawasaki
  - Kobe University Hospital, Kobe
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Dokkyo Medical University Saitama Medical Center, Minamikoshigaya
  - Nagasaki University Hospital, Nagasaki
  - Nagoya City University Hospital, Nagoya
  - Kochi Medical School Hospital, Nankoku
  - Niigata University Medical and Dental Hospital, Niigata
  - National Hospital Organization Okayama Medical Center, Okayama
  - Tohoku University Hospital, Sendai
  - Ntt Medical Center Tokyo, Shinagawa-ku
  - Tokyo Medical University Hospital, Shinjuku-ku
  - Osaka University Hospital, Suita
  - National University Corporation - Tokyo Medical and Dental University (Tmdu), Tokyo
  - Juntendo University Urayasu Hospital, Urayasu
  - Yamagata University Hospital, Yamagata
- Mexico (6):
  - Trials in Medicine S.C., Deleg. Cuauhtemoc
  - Instituto de Investigaciones Aplicadas A La Neurociencia A.C, Durango
  - Centro de Dermatologia de Monterrey, Monterrey
  - Universidad Autonoma de Nuevo Leon (Uanl) - Hospital Universitario Dr. Jose Eleuterio Gonzalez - Cen, Monterrey
  - Clinica de Enfermedades Cronicas Y de Procedimientos Especiales (Cecype), Morelia
  - Grupo Clínico Catei Sc, Providencia 5TA Seccion
- Netherlands (2):
  - Uva - Amc - Stichting Nederlands Instituut Voor Pigmentstoornissen (Snip) (Netherlands Institute For, Amsterdam
  - Bravis Ziekenhuis, Bergen op Zoom
- Poland (13):
  - Dermapolis Medical Dermatology Center Dr N. Med. Edyta Gebska, Chorzów
  - Synexus Polska Sp Z Oo Oddzial W Czestochowie, Częstochowa
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Synexus Polska Sp. Z O.O. Oddzial W Katowicach, Katowice
  - Synexus Polska Sp Z Oo Oddzial W Lodzi, Lodz
  - Dermodent Centrum Medyczne Aldona Czajkowska Rafa¿ Czajkowski, Osielsko
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski
  - Uniwersytecki Szpital Kliniczny Im. Fryderyka Chopina W Rzeszowie, Rzeszów
  - Panstwowy Instytut Medyczny Mswia, Warsaw
  - Carpe Diem Centrum Medycyny Estetycznej, Warsaw
  - Synexus Polska Sp. Z O.O. Oddzial W Warszawie, Warsaw
  - Etg Warszawa, Warsaw
  - Emc Instytut Medyczny Spolka Akcyjna-Euromedicare Szpital Specjalistyczny Z Przychodnia, Wrocaw
- Spain (6):
  - Hospital Universitario Fundacion Alcorcon, Alcorcón
  - Hospital Universitari Germans Trias I Pujol (Hugtp), Badalona
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Clinica Universidad de Navarra (Cun), Madrid
  - Hospital de Manises, Manises

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A study to Evaluate Efficacy and Safety of Povorcitinib in Participants With Nonsegmental Vitiligo (STOP-V1) — https://www.incyteclinicaltrials.com/study/?id=INCB54707-303&SearchTerm=INCB54707-303&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=